CLINICAL TRIAL: NCT04636125
Title: Prospective Evaluation of Oral Antibiotics for Treatment of Shoulder PJI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNAM18D.443
Record Dates: First submitted 2020-10-21; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Periprosthetic Infection; Oral Antibiotics; Revision Total Shoulder Arthroplasty
MeSH Terms: interventions — Doxycycline; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Revision Total Shoulder Arthroplasty (Other): Routine cultures are taken at the time of surgery. All patients are seen by an Infectious Disease Specialist and placed on 2 weeks oral doxycycline 100 mg (or alternative based on allergy or sensitivity) pending culture results.
  Interventions: Drug: Doxycycline 100 MG Oral Tablet

INTERVENTIONS:
Drug: Doxycycline 100 MG Oral Tablet — Patients that are undergoing a single stage revision total shoulder arthroplasty will be enrolled in this study. As is standard of care, routine cultures will be taken from predetermined areas in the shoulder. All patients will be treated with 13 days of oral Doxycycline pending culture results.

SUMMARY:
Cutibacterium acnes (C. acnes) is an anaerobic aerotolerant bacteria commonly isolated during revision shoulder surgery. It is increasingly recognized as a pathogen, mainly in implant-related infections. As an anaerobe, it usually needs a prolonged culture incubation time of up to 14 days for growth and the association between implant surgery and C. acnes infection is not always obvious. Unfortunately, prolonged incubation also increases the risk of false positive cultures in isolating organisms that may exist as a result of contamination. Given high rates of positive C. acnes cultures in cases of both primary and revision shoulder surgery, the ramifications of positive C. acnes cultures for clinical decision making remains uncertain.

The purpose of this study is to prospectively study the efficacy and side-effect profile of surgical treatment plus an oral antibiotic regiment for shoulder PJI with indolent organisms (C. acnes and CNS).

ELIGIBILITY:
Inclusion Criteria:

1. all patients undergoing single-stage revision arthroplasty with all implants exchanged,
2. all patients undergoing single-stage revision arthroplasty with some implants retained,
3. all patients undergoing explantation of a shoulder arthroplasty and placement of an antibiotic spacer

Exclusion Criteria:

1. patients with polymicrobial infection,
2. patients with infection by organisms other than P. acnes or Coagulase Negative Staphylococcus,
3. patients with clinical suspicion of infection but negative cultures,
4. patients with no preoperative or intraoperative signs of infection and only 1 positive culture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-09-24 (Estimated); Study Completion 2021-09-24 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Infections | 1 year
  The investigator will measure the incidence of postoperative infections in participants treated with oral antibiotics after revision shoulder surgery versus those treated with intravenous antibiotics after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States